CLINICAL TRIAL: NCT04624984
Title: PD-1 Inhibitor or PD-1 Inhibitor Plus GVD(Gemcitabine, Vinorelbine and Doxorubicin Liposome) Regimen for Relapsed/Refractory Classical Hodgkin Lymphoma (R/R CHL): a Single Arm, Open Label, Phase II Study
Brief Title: PD-1 Inhibitor or PD-1 Inhibitor Plus GVD for Relapsed/Refractory CHL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-238-01
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Classical Hodgkin Lymphoma; Refractory or Relapsed Classical Hodgkin Lymphoma
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Gemcitabine; Vinorelbine; Doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 Inhibitor or PD-1 Inhibitor with GVD (Experimental): All patients receive PD-1 Inhibitor on day 1. Treatment cycles repeat every 3 weeks for 3 cycles in the absence of disease progression or unacceptable toxicity. Patients with PET/CT confirmed CR or PR receive PD-1 Inhibitor for another 3 cycles. Patients with PD or SD receive PD-1 Inhibitor plus GVD (gemcitabine, vinorelbine and doxorubicin liposome) regimen every 3 weeks for up to 4 cycles in the absence of disease progression or unacceptable toxicity.
  Patients with PET/CT confirmed CR after 6 cycles of PD-1 Inhibitor treatment can receive radiotherapy or ASCT, which is determined by investigators. Patients with PR receive 2-4 cycles of PD-1 Inhibitor plus GVD regimen. Patients with PD or SD receive 4 cycles of PD-1 Inhibitor plus GVD regimen.
  Patients with confirmed CR or PR after PD-1 Inhibitor plus GVD regimen can receive radiotherapy or ASCT, which is determined by investigators. Patients with PD or SD quit the trial.
  Interventions: Drug: PD-1 inhibitor; Drug: PD-1 inhibitor, gemcitabine, vinorelbine and doxorubicin liposome

INTERVENTIONS:
Drug: PD-1 inhibitor — PD-1 Inhibitor, intravenous drip, d1.
Drug: PD-1 inhibitor, gemcitabine, vinorelbine and doxorubicin liposome — PD-1 Inhibitor, intravenous drip, d1; Gemcitabine, 1000mg/m2, intravenous drip, d1,d8; Vinorelbine, 50mg/m2, PO, d1,d8; Doxorubicin Liposome, 30mg/m2, intravenous drip, d1;

SUMMARY:
This phase 2 trial studies the efficacy and safety of PD-1 inhibitor monotherapy or PD-1 inhibitor with GVD (Gemcitabine, Vinorelbine and Doxorubicin Liposome) regimen for relapsed or refractory classical Hodgkin lymphoma (CHL) patients who failed the first-line induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed classical Hodgkin lymphoma;
* Refractory to or relapsed after first-line induction therapy; prior radiotherapy is allowed;
* At least one evaluable lesion according to 2014 Lugano criteria;
* Life expectancy > 3 months;
* Eastern Cooperative Oncology Group (ECOG) of 0-1;
* Able to participate in all required study procedures;
* Proper functioning of the major organs: 1) The absolute value of neutrophils (>1.5×10^9/L); 2) platelet count (> 75×10^9/L); 3) Hemoglobin (> 80 g/L); 4) Serum creatinine <1.5 times Upper Limit Normal (ULN) ; 5) Serum total bilirubin < 1.5 times ULN; 6) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) < 2.5 times ULN; 7) Coagulation function: International Normalized Ratio (INR), Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) < 1.5 times ULN (unless the subject is receiving anticoagulant therapy and PT and APTT are within the expected range at screening time). ; 8) Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (±10%);
* There was no evidence that subjects had difficulty breathing at rest, and the measured value of pulse oximetry at rest was more than 92%;
* Volunteers who signed informed consent.

Exclusion Criteria:

* Involvement of central nervous system (CNS);
* Previously received treatment of immune checkpoint inhibitors (eg. PD-1, PD-L1, CTLA-4);
* Previously received treatment of hematopoietic cell transplantation;
* Patients with Hemophagocytic syndrome;
* Patients with active autoimmune diseases requiring systematic treatment in the past two years (hormone replacement therapy is not considered systematic treatment, such as type I diabetes mellitus, hypothyroidism requiring only thyroxine replacement therapy, adrenocortical dysfunction or pituitary dysfunction requiring only physiological doses of glucocorticoid replacement therapy); Patients with autoimmune diseases who do not require systematic treatment within two years can be enrolled;
* Requiring treatment with corticosteroids or other immunosuppressive drugs within 14 days of study drug administration [allowing subjects to use local, ocular, intra-articular, intranasal and inhaled glucocorticoid therapy (with very low systemic absorption); and allowing short-term (< 7 days) glucocorticoid prophylaxis (e.g., contrast agent overdose sensitivity) or for the treatment of non-autoimmune diseases (e.g. delayed hypersensitivity caused by contact allergens).
* Uncontrolled active infection, with the exception of tumor-related B symptom fever;
* History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome are known;
* Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA (no more than 10^4 copies/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 10^4 copies/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group;
* Diagnosed with or receiving treatment for malignancy other than lymphoma;
* Pregnant or breastfeeding women;
* Other researchers consider it unsuitable for patients to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 2 years
  Complete remission rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Objective Response rate | 2 years
  Objective Response rate will be determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression Free Survival | 5 years
  The time from the start of treatment to the progression of the tumor or death (due to any cause).
Overall Survival | 5 years
  The time from the start of treatment to time of death (due to any cause).
Duration of Response | 5 years
  The time from the first assessment of complete remission or partial remission to progressive disease or death (due to any cause).
Time to Response (TTR) | 2 years
  The time from the start of treatment to the first assessment of complete remission or partial remission.
Percentage of Participants With Adverse Events | 2 years
  Adverse Events will be determined and graded on the basis of investigator assessments according to NCI CTC AE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Qingqing Cai, MD, Principal Investigator — Sun Yat-sen University
Locations (3):
- China (3):
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University,, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University, Guangzhou, Guangdong